CLINICAL TRIAL: NCT05025436
Title: Laser Acupuncture Improves Constipation for Critical Care Nurses During the COVlD-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hui-Yu Lin (Other)
Responsible Party: Sponsor-Investigator, Hui-Yu Lin, Nurse, Far Eastern Memorial Hospital
Organization: Far Eastern Memorial Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 109156-F
Record Dates: First submitted 2021-07-28; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Nurse
Keywords: Laser pointer; constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: The intervention time of the study was 2.5 months. The cross-over test was adopted. There were 2 kinds of intervention measures. Each subject in the experimental group was given the main acupoints (5 acupoints) and the physical acupoints (1-2 acupuncture points). Acupoints) Intervene in low-energy laser (Erger laser pen) acupoint stimulation, set wavelength 810nm +/-10%, power 200mW, select Bahr parameter (B2: 1199 Hz; B3: 2398 Hz) module according to the acupuncture point for treatment The time is 30 seconds per acupoint, and the therapeutic dose is 3 joules per acupoint; each subject in the control group is given the same main acupoints and physical matching acupoints without energy acupoint care (therapeutic dose is 0 joules per acupoint), three times a week, for a period of 4 Weeks later, after a 2-week suspension, the two groups crossed over for another 4 weeks of intervention.
Who Masked: Participant
Masking Description: A total of 64 subjects were admitted, and they were randomly assigned into a control group and an experimental group by a crossover test, with 32 persons in each group. Random Allocation Software is used to randomly allocate 64 cases with random serial numbers generated by the computer. The 64 cases are divided into two groups with 32 people in each group. Randomly assigned serial numbers will be stored in consecutively numbered opaque sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupoint Laser Group (Experimental): Each subject in the experimental group was given the same main acupoints (5 acupoints) and physique matching acupoints (1-2 acupoints) interventional low-energy laser (Erger laser pen) acupoint stimulation, set wavelength 810nm +/- 10%, power 200mW, select Bahr parameter (B2: 1199 Hz; B3: 2398 Hz) module according to acupoints, treatment time is 30 seconds per acupoint, and the treatment dose is 3 joules per acupoint three times a week. After a period of 4 weeks, pause 2 After two weeks, the two groups crossed over and carried out 4 weeks of intervention.
  Interventions: Device: Acupoint stimulation with low energy laser (Erger laser pen)
- Control Group (No Intervention): Each subject in the control group was given the same main acupoints (5 acupoints) and constitution matching acupoints (1-2 acupoints) without energy acupoint care (therapeutic dose is 0 joules per acupoint), three times a week, after 4 weeks After a two-week suspension, the two groups crossed over for another four-week intervention.

INTERVENTIONS:
Device: Acupoint stimulation with low energy laser (Erger laser pen) — Each subject was given the same main acupoints (5 acupoints) and physique matching acupoints (1-2 acupoints) interventional low-energy laser (Erger laser pen) acupoint stimulation, set wavelength 810nm +/-10%, The power is 200mW, and the Bahr parameter (B2: 1199 Hz; B3: 2398 Hz) module is selected according to the acupoints. The treatment time is 30 seconds per acupoint, and the treatment dose is 3 joules per acupoint three times a week. After a period of 4 weeks, after a 2-week pause, After the two groups crossed for 4 weeks, each subject was given the same main acupoints (5 acupoints) and physique matching acupoints (1-2 acupoints) with low-energy laser (Erjie laser pen) acupoint stimulation. Set wavelength 810nm +/-10%, power 200mW, select Bahr parameter (B2: 1199 Hz; B3: 2398 Hz) module according to acupoints, treatment time is 30 seconds per acupoint, and treatment dose is 3 joules per acupoint three times a week for a period of time 4 weeks.
  Arms: Acupoint Laser Group

SUMMARY:
According to the "Survey on Colon Pouch Problems and Living Settlements" conducted by the Taiwan Cancer Foundation in 2017, 48% of office workers have constipation problems. The proportion of medical staff is high, especially in acute and severe units. The reason is high work pressure. , Life tension and other characteristics. In western medicine, enemas or stool softening drugs are often used in clinical treatment. This kind of treatment treats the symptoms but not the root cause. In addition, long-term use can easily cause damage to the intestinal nerves and become dependent on drugs. Systematic literature points out that the use of acupoint stimulation can effectively increase spontaneous defecation and promote bowel movements, but there is no conclusion on the effective acupuncture points. Therefore, the purpose of this research is to use precise acupoint stimulation to improve the constipation problem of nursing staff in emergency and intensive care units.

This study adopts a single-blind randomized controlled Cross-over trial. Take the emergency department of a medical center in the north as the research site, and take the nursing staff of the emergency and intensive care unit with constipation as the research object. The experimental group received precise acupoint care, and the control group received routine care. After a 2-week pause, the two groups crossed. Use questionnaires to collect basic patient data (basic attributes and Chinese medical physique, etc.), and assess the intestinal tract. Data analysis uses IBM SPSS 22.0 software for descriptive statistical analysis and inferential statistical analysis, and p<0.05 is regarded as statistically significant.

DETAILED DESCRIPTION:
1. Research purpose:

1. Explore the effect of acupoint stimulation on constipation of emergency and intensive nursing staff.
2. Explore the effect of acupoint stimulation on bowel movements of nursing staff in acute and intensive care.
3. Explore the effect of acupoint stimulation on the quality of life of emergency and intensive nursing staff.

2. Research methods:

1. Selection criteria and number of people.

   1. Number of subjects accepted: _64_ people in this hospital, _0_ people in other centers A total of 64 people were admitted to the Yadong Memorial Hospital, and they were randomly assigned to a control group and an experimental group by a crossover test, with 32 people in each group.
   2. Conditions of inclusion:

      1. Over 20 years old.
      2. Emergency nursing staff with constipation.
      3. Willing to participate in this research and sign a consent form.
   3. Exclusion conditions:

      1. Nursing staff with organic disease.
      2. Nursing staff with a history of gastrointestinal surgery.
      3. Nursing staff with intestinal adhesions.
      4. Nursing staff with a cardiac rhythm device.
      5. Nursing staff with abdominal tumors.
      6. Pregnant nursing staff.
   4. Recruitment method:

      This study is expected to target emergency nurses with constipation in the emergency department of Yadong Memorial Hospital. The co-host will use 5-10 minutes in the emergency nurse handover meeting to announce the research topic "The effectiveness of precision acupoint care on constipation improvement of nurses in emergency and intensive care units". If there are suitable subjects, they will first ask if they are willing to participate in this research. With the consent of the subjects, the co-host of the project will make an appointment with the subjects in the emergency meeting room, and explain the purpose, procedures, process and emergency treatment process face to face.
   5. Method of consent of research subjects:

      1. The co-host of the project, Lin Huiyu, the nurse manager, learned of the willing subjects in the emergency department and informed the host of the project by telephone. The co-host of the project made an appointment with the subjects in the emergency meeting room and explained the research process face to face. For related matters, a consent form will be given to the signed subjects.
      2. Let the subjects understand the purpose of the research and the process and methods of collecting data. If the subjects feel uncomfortable during the research process, they can withdraw and terminate the research at any time without affecting their original treatment and care. Treatment methods to improve constipation, such as enema, medication, diet, etc.).
2. Research design:

   1. Method of research:

      This research plan applies for the approval of the Human Test Review Committee of Yadong Memorial Hospital and the relevant departments or units of the hospital to start accepting the case. It is estimated that emergency nurses with constipation symptoms will be the research subjects, and the number of samples to be collected will be estimated through G-power version 3.1 statistical software, and a total of 64 people (32 people in each group) will be included. Random Allocation Software is used to randomly allocate 64 cases with random serial numbers generated by the computer. The 64 cases are divided into two groups with 32 people in each group. Randomly assigned serial numbers will be stored in consecutively numbered opaque sealed envelopes.

      On the first day of admission, the host/co-host will explain the case acceptance and research progress in the emergency meeting room, and complete basic information and pre-test questionnaires. It takes 13 minutes. The intervention time of the study was 2.5 months. The method of cross-over was adopted. There were 2 kinds of intervention measures. Each subject in the experimental group was involved in acupoint stimulation with a low-energy laser (Erger laser pen), and set Wavelength 810nm +/-10%, power 200mW, select Bahr parameter (B2: 1199 Hz; B3: 2398 Hz) module according to acupoints, treatment time is 30 seconds per acupoint, treatment dose is 3 joules per acupoint, select main acupoint as day Shu points, Zusanli points, Hegu points, Zhigou points, Shangjuxu points, and physique matching points: the physique matching point for yang deficiency is Zhaohai; the yin deficiency physique matching point is Sanyinjiao and Taixi points; the qi deficiency constitution matching point is There are Fenglong and Sanyinjiao points; Quchi is the matching point for physical heat (dampness and heat, phlegm-dampness); Yanglingquan is the matching point for Qi stagnation (qi stagnation and blood stasis); each of the control group Subjects were given the same main acupoints (5 acupoints) and physical matching acupoints (1-2 acupoints) without energy acupoint care (therapeutic dose is 0 joules per acupoint), three times a week, after a period of 4 weeks, pause for 2 weeks Later, after the two groups crossed, interventional measures were carried out for 4 weeks. The measurement time and method are: Bristol stool classification table, visual analogy scale for constipation symptoms, bowel movement, constipation assessment scale, and Chinese version of the patient constipation symptom scale on the day of admission (before intervention). , Chinese medicine body mass scale, Chinese version of self-rating quality of life for patients with constipation scale, Chinese version of Bayesian Anxiety Scale, and Bristol Stool Classification Scale and Visual Analogy Scale for Constipation Symptoms to investigate stool status (one week) 3 times), and auscultation for 1 minute before and after each intervention to investigate the stool status. After the intervention, the constipation assessment scale will be measured once a week after the intervention, and the Chinese version of the patient constipation symptom scale will be conducted every two weeks, the fourth week After the interventional measures are completed, the TCM body mass scale, the Chinese version of the Bayesian Anxiety Scale, and the Chinese version of the self-assessment of the quality of life for patients with constipation will be tested. It takes 10 minutes to complete the post-test questionnaire.
   2. Subject tracking or necessary rehabilitation plan:

      During the study, closely follow up and pay attention to whether the subjects have the following discomforts: skin rashes at the acupoints, abnormal skin sensations, fatigue, slight dizziness and other symptoms. If the above symptoms occur, immediately stop the low-energy laser Shot pen) acupoint stimulation.
   3. Treatment effect evaluation and statistical analysis methods:

The researcher first checks the integrity of the data, encodes the data, and then enters it into the computer according to the codebook. After the file is created, the IBM SPSS 22.0 software is used for statistical analysis of the data. In this study, p<0.05 was regarded as statistically significant. According to the purpose of the research and the nature of the variables, the following statistical methods are used for descriptive statistical analysis and inferential statistical analysis. Descriptive statistical analysis: categorical variables are described by sample number, percentage, and chi-square test, while continuous variables are described by average, standard deviation, and independent sample t test; inferential statistical analysis: Generalized Estimating Equations (GEE) ): Analyze the correlation between repeated measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Be over twenty years old.
2. Emergency nursing staff with constipation.
3. Willing to participate in this research and sign a consent form.

Exclusion Criteria:

1. Nursing staff with organic disease.
2. Nursing staff with a history of gastrointestinal surgery.
3. Nursing staff with intestinal adhesions.
4. Nursing staff with a cardiac rhythm device.
5. Nursing staff with abdominal tumors.
6. Pregnant nursing staff.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
To explore the effect of acupoint stimulation on constipation of emergency and intensive nursing staff. | 2.5 months.
  Use patient assessment of constipation symptom (PAC-SYM) with a minimum score of 0 and a maximum of 48. The higher the score, the more serious the constipation; the constipation assessment scale (CAS), the minimum is 0 and the maximum is 16, the higher the score, the more severe the constipation; The Bristol Stool Scale is divided into types 1 to 7, the first type is severe constipation, and the seventh type is severe diarrhea. The score is evaluated every day to understand the subject's constipation.
To explore the effect of acupoint stimulation on bowel movements of nursing staff in acute and intensive care. | 2.5 months.
  Before and after each acupoint stimulation, auscultate the subject's bowel movements to evaluate the increase in the number of bowel movements.
To explore the effect of acupoint stimulation on the quality of life of nursing staff in acute and intensive care. | 2.5 months.
  Use Patient Assessment of Constipation Quality of Life (PAC-QOL) to evaluate the quality of life of patients with constipation. The lowest score is 0 and the highest is 112. The higher the score, the worse the quality of life caused by constipation.

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei County, Taiwan